CLINICAL TRIAL: NCT05236244
Title: Does the Effect of Mental Fatigue Created by Motor Imagery on Upper Extremity Functions Change With Diaphragmatic Breathing Exercises
Brief Title: Motor Imagery in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bandırma Onyedi Eylül University (Other)
Responsible Party: Principal Investigator, Burçin Akçay, Assistant Professor, Bandırma Onyedi Eylül University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BurcinAkcay
Record Dates: First submitted 2022-02-02; First posted 2022-02-11 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Health, Subjective
Keywords: motor imagery; mental fatigue; diaphragmatic breathing exercises
MeSH Terms: conditions — Mental Fatigue

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- İntervention group (Experimental): Diaphragmatic breathing exercises: First Evaluation + (1 week break) + Motor imagery protocol + Second Evaluation + 8 weeks of diaphragmatic breathing exercises +Third Evaluation +(1 week interval) + Motor imagery protocol + Fourth Evaluation
  Interventions: Other: İntervention group
- Control Group (No Intervention): First Evaluation + (1 week break) + Motor imagery protocol + Second Evaluation + 8 weeks break +Third Evaluation +(1 week interval) + Motor imagery protocol + Fourth Evaluation

INTERVENTIONS:
Other: İntervention group — Diaphragmatic Breathing Exercises
  Arms: İntervention group

SUMMARY:
The research will be the first to examine the relationship between mental fatigue induced by motor imagery and upper extremity performance. This study, it is aimed to examine whether the effects of mental fatigue created by motor imagery on upper extremity performance can be reduced by diaphragmatic breathing exercises.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed dominance (it will be decided according to Edinburgh Hand Questionnaire Result)
* Volunteer to participate in the study.
* To be sedentary
* Not having any problems that prevent breathing exercises
* Be between the ages of 18-30

Exclusion Criteria:

* Have any mental or sensory problems in the past 6 months
* Presence of acute infection or chronic disease of neurological, psychiatric, orthopedic, cardiological, rheumatological, etc.
* Having had Covid-19
* Having any respiratory disease (asthma, COPD, etc.)
* Having any upper extremity injury and/or operation (trauma, surgery, fracture, etc.) in the -Last 6 months doing regular exercises (at least 30 minutes a day / 5 times a week for a total of at least 150 minutes)
* Be on regular medication
* Be smoking

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
1-Isometric Elbow Flexion Force | 8 weeks
  1-Isometric Elbow Flexion Force: The participant will try to move their hands towards their shoulder as forcefully as possible for 2-3 seconds with their upper arms at their sides, elbow bent at 90 degrees and forearm in supination.
2-Handgrip strength | 8 weeks
  2-Handgrip strength: Handgrip strength will be assessed using a Jamar hand dynamometer (Lafayette Instrument Company, USA).
3-Upper extremity reaction test | 8 weeks
  3-Upper extremity reaction test: It is planned to use a validated BlazePod sensor for upper extremity reaction time test
4-Finger reaction test | 8 weeks
  4-Finger reaction test: By placing the dominant hand index finger on the left button of a computer mouse, the participant will be asked to press the left button as soon as the traffic light pattern glows green on the screen.
5-Hand performance test | 8 weeks
  5-Hand performance test: A nine-hole peg test will be used.
6-Position Sense | 8 weeks
  6-Position Sense: The height of the laser track marker test target board can be adjusted according to the height of the person, and the zero point will be aligned for each patient's glenohumeral joint separately. A standardized coordinate system drawn on the target board will show the different angles of motion calculated using a formula.
7-Tactile sense | 8 weeks
  7-Tactile sense: The calibrated Semmes Weinstein monofilament test (North Coast Medical, USA) will be used to measure perceptual thresholds for cutaneous stimuli (Bell-Krotoski, Fess, Figarola, & Hiltz, 1995; Dannenbaum, Michaelsen, Desrosiers, & Levin, 2002).
8-Two-point discrimination | 8 weeks
  8-Two-point discrimination: The two-point discrimination test is the evaluation of the ability to detect stimuli applied from two different points at the same time.
9-Upper extremity endurance test | 8 weeks
  9-Upper extremity endurance test: After weighing the body weight, the weight to be held in the hand will be calculated as 2% of the body weight and if it is fractional, it will be rounded to the nearest 0.5 kg. The participant will hang the test arm out of the bed. Here he has to take the weight in his hand and raise it so that the "thumb faces up" and the arm is 90° horizontally. A metronome set to 60 Hz will then be used to standardize the test; in this way, participants will be instructed to raise their arms at the first beep, to keep the arm in 90 abduction during the next beep, and then to lower them to the starting position with the third beep. The test will be terminated as a result of fulfilling any of the following termination criteria (Moore, Uhl, & Kibler, 2013).

SECONDARY OUTCOMES:
Mental Fatigue (VAS) | 8 weeks
  VAS: In our study, mental fatigue level will be evaluated with VAS. VAS is a valid and reliable method for measuring the severity of fatigue and is a one-dimensional scale widely used in the clinic. In practice, patients are asked to choose the number that best describes the severity of fatigue they feel. Zero means not tired, 10 means very tired.

CONTACTS AND LOCATIONS:
Locations (1):
- BandırmaOnyediEylulU, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No